CLINICAL TRIAL: NCT05873725
Title: Retrospective Study of High Dose Follitropin Delta in a Mixed Protocol With Human Chorionic Gonadotropin
Acronym: STORM
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3282
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: IVF; Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin delta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Follitropin delta + hCG: Combination of follitropin delta and serial hCG injections at individualized doses, where dosing regimen was determined according to AMH and weight in women undergoing an IVF antagonist cycle
  Interventions: Drug: Follitropin delta
- Follitropin delta + HP-hMG: Combination of follitropin delta and highly-purified human menopausal gonadotropin (HP-hMG) where dosing regimen was determined according to AMH and weight in women undergoing an IVF antagonist cycle
  Interventions: Drug: Follitropin delta

INTERVENTIONS:
Drug: Follitropin delta — Evaluation of the IVF cycle using the prescribed medication

SUMMARY:
Follitropin delta is a rFSH, uniquely expressed in a human fetal retinal cell line, which owing to differences in glycosylation profile has a lower clearance and induces a higher ovarian response in humans than existing rFSH preparations when administered at equal doses of biological activity. A noninferiority clinical trial (ESTHER-1) in which individualized dosage of follitropin delta according to each patient's profile (AMH and weight) was compared to conventional follitropin alfa dosing for IVF have demonstrated that an individualized follitropin delta dosing is noninferior to conventional follitropin alfa with respect to ongoing pregnancy rate, ongoing implantation rate, and also live births, with a concomitant reduction in iatrogenic complications, including OHSS

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 42 years of age undergoing IVF/ICSI cycle
* IVF antagonist protocol
* Regular menstrual cycles of 24-35 days
* Presence of both ovaries

Exclusion Criteria:

* Endometriosis stage III/IV
* History of recurrent miscarriages, defined as ≥ 3 consecutive losses
* Women undergoing ovarian stimulation for oncologic or elective fertility preservation
* Women participating in any other research project
* Hypersensitivity to follitropin delta and/or human chorionic gonadotropin
* Use of Growth Hormone (GH) during the stimulation cycle

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Women consulting the clinic for fertility issues that require in vitro fertilization
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Number of good quality blastocysts | Up to 6 day
  Number of good quality oocytes fertilized

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada